CLINICAL TRIAL: NCT04005313
Title: Development and Application of Portable Multisensory Stimulation Device: Vibroacustic Therapy
Brief Title: Development and Application of Portable Multisensory Stimulation Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB105-116-A; 107-2218-E-320 -001 - (Other Grant/Funding Number: Ministry of science and technology); 106-2218-E-320 -001 - (Other Grant/Funding Number: Ministry of science and technology); IRB107-39-B (Other: Buddhist Tzu Chi Hospital)
Record Dates: First submitted 2019-05-30; First posted 2019-07-02 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Cognitive Impairment
Keywords: Electromyographic activity; Neck pain; Electroencephalographic activity; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Neck Pain; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Comparison between unisensory and multisensory stimulation (Experimental): The same person receive unisensory and multisensory stimulation on separate day.
  Interventions: Device: vibroacoustic device
- The treatment effect of multisensory stimulation (Experimental): The persons living in long-term care facility would receive multisensory stimulation for one month.
  Interventions: Device: vibroacoustic device
- Multisensory stimulation and virtual reality. (Experimental): The subjects would receive vibroacoustic therapy or virtual reality.
  Interventions: Device: vibroacoustic device
- Vibroacustic therapy on neck pain. (Experimental): The subjects would receive either vibroacustic therapy or music therapy.
  Interventions: Device: vibroacoustic device

INTERVENTIONS:
Device: vibroacoustic device — the participants will receive the vibroacustic device or music therapy

SUMMARY:
This is a study to develop the vibroacustic devices, and to compare the effects between vibroacustic device therapy and music therapy in adults with dementia or with neck pain. The immediate effect and long-term training effect would be assessed.

DETAILED DESCRIPTION:
The outcome measures included functional assessment ( such as: range of motion, balance etc.) and neurolphysiological assessment (such as: electroencephalographic activity or electromyographic activity).

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate Dementia
* age-matched healthy subjects

Exclusion Criteria:

* can not follow order

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
the electroencephalographic (EEG) activities ncluding Alpha, Beta, Theta, and Delta signals will be assessed in persons with mild to moderate dementia and healthy subjects.after sensory stimulation. . | one year
  The EEG was recorded by EMOTIV EPOC+ mobile headset (Bioinformatics Company, USA). The wireless 14-EEG channels on the skull were located at anterior frontal (AF), frontal (F), frontal central (FC), temporal (T), parietal (P) and occipital (O) areas,The frequency analysis of brain waves includinh Alpha, Beta, Theta, and Delta signals before, during and after sensory stimulation will be recorded and analyzed.

SECONDARY OUTCOMES:
The pressure pain threshold following multisensory stimulation will be assessed around cervical region. | one year
  The pressure pain threshold was measured by MicroFET3 ( Hoggan Health Industries, Utah, USA) at cervical region including cervical erector (CE), upper trapezius (UT) and sternocleidomastoid (SCM). At the trigger point of the muscle, the pressure of the test group is increased at a rate of about 1 newton/second. When the subject feels uncomfortable, the active stop is the end point of the test for perceived pain threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Chich-Haung Yang, PhD, Principal Investigator — Tzu Chi University
Locations (1):
- Kwan-Hwa Lin, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beinert K, Englert V, Taube W. After-effects of neck muscle vibration on sensorimotor function and pain in neck pain patients and healthy controls - a case-control study. Disabil Rehabil. 2019 Aug;41(16):1906-1913. doi: 10.1080/09638288.2018.1451925. Epub 2018 Mar 21. PMID 29558836